CLINICAL TRIAL: NCT01759901
Title: Open Liver Resection With or Without Vascular Inflow Occlusion for Hepatocellular Carcinoma: a Randomized Controlled Trial
Brief Title: Effect of Vascular Inflow Occlusion in Open Liver Resection for Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Yue Sun, Clinical Assistant Professor (honorary), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2012.351-T
Record Dates: First submitted 2013-01-01; First posted 2013-01-03 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatectomy; vascular inflow occlusion
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pringle (Experimental): Intermittent vascular inflow occlusion applied during liver resection
  Interventions: Procedure: Pringle
- Non-Pringle (No Intervention): No vascular inflow occlusion applied during liver resection

INTERVENTIONS:
Procedure: Pringle — Vascular clamp is applied across hepatoduodenal ligament intermittently in 15 minutes on / 5 minutes off interval
  Other Names: Vascular inflow occlusion
  Arms: Pringle

SUMMARY:
Bleeding is a major problem during liver resection. Vascular inflow occlusion, also known as Pringle maneuver, has been commonly employed to reduce blood loss during liver surgery. However, Pringle maneuver might cause ischaemic insult to the remnant liver and lead to post-operative liver dysfunction.

The investigators hypothesize that liver resection without the use of vascular inflow occlusion (Pringle maneuver) is associated with lower postoperative complications rate.

The aim of this study is to evaluate whether elective open liver resection without vascular inflow occlusion (Pringle Maneuvre) would lead to a reduction of post-operative surgical complications in patient with hepatocellular carcinoma.

Eligible patients undergoing liver resection in the Prince of Wales Hospital will be recruited and randomized into 2 study arms comparing the effect of Pringle maneuver.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Child's A or B cirrhosis

Exclusion Criteria:

* Informed consent not available
* Presence of portal vein thrombosis, portal vein tumor thrombus, or previous portal vein embolisation
* Presence of hepatic artery thrombosis, previous transarterial therapy like TACE, lipiodol-ethanol mixture injection or transarterial internal radiation
* Anticipation of portal vein resection
* Emergency hepatectomy
* Ruptured HCC
* Adhesion or anatomical variation that preclude safe and successful application of Pringle maneuver
* Anticipation of concomitant bowel or bile duct resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Post-operative surgical complications | 1 month
  30-day morbidity after open liver resection, which includes ascites, pleural effusion, wound infection and intra-abdominal collection

SECONDARY OUTCOMES:
Other post-operative complications | 1 month
  post-operative liver failure, post-op mortality, operative blood loss, duration of operation and hospital stay
Survival | 5 year
  Overall and disease-free survival at 1, 3, 5-year
Recurrence rate of hepatocellular carcinoma | 5 year
  Recurrence rate of hepatocellular carcinoma at 1,3,5 year

CONTACTS AND LOCATIONS:
Overall Officials: Kit Fai Lee, MBBS, Principal Investigator — Clinical Associate Professor (honorary)
Locations (1):
- The Prince of Wales Hospital, Hong Kong, China

REFERENCES:
- [Derived] Lee KF, Chong CCN, Cheung SYS, Wong J, Fung AKY, Lok HT, Lai PBS. Impact of Intermittent Pringle Maneuver on Long-Term Survival After Hepatectomy for Hepatocellular Carcinoma: Result from Two Combined Randomized Controlled Trials. World J Surg. 2019 Dec;43(12):3101-3109. doi: 10.1007/s00268-019-05130-8. PMID 31420724
- [Derived] Lee KF, Wong J, Cheung SYS, Chong CCN, Hui JWY, Leung VYF, Yu SCH, Lai PBS. Does Intermittent Pringle Maneuver Increase Postoperative Complications After Hepatectomy for Hepatocellular Carcinoma? A Randomized Controlled Trial. World J Surg. 2018 Oct;42(10):3302-3311. doi: 10.1007/s00268-018-4637-3. PMID 29696328